CLINICAL TRIAL: NCT04717908
Title: Refining MDR-TB Treatment (T) Regimens (R) for Ultra(U) Short(S) Therapy(T) (TB-TRUST)-PLUS
Brief Title: Refining MDR-TB Treatment (T) Regimens (R) for Ultra(U) Short(S) Therapy(T)-PLUS
Acronym: TB-TRUSTplus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY1214
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Multidrug resistant tuberculosis; shorter treatment; all-oral regimen; PZA sensitivity
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — bedaquiline; Pyrazinamide; Linezolid; Cycloserine; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PZA sensitivity guided all oral regimen (Experimental): This regimen consists of two periods of 24-36 weeks. During the first 4-8 weeks(waiting for pyrazinamide drug sensitivity test), the regimen consists of bedaquiline, linezolid, cycloserine, clofazimine and pyrazinamide. Then based on molecular PZA drug sensitivity results, patients will be divided into three sub-groups.
  The regimen for PZA-S patients, consisting of bedaquiline, linezolid, cycloserine and pyrazinamide, are given until the 24th week (prolonged to 28 or 32 weeks if no smear conversion by end of 16th and 20th week).
  PZA-R sub-group regimen, consisting of bedaquiline, linezolid, cycloserine and clofazimine ,are given until 36th week (prolonged to 40 or 44 weeks if no smear conversion by end of 16th and 20th week) .
  PZA-U sub-group continue the previous regimen, consisting of bedaquiline, linezolid, cycloserine , clofazimine and pyrazinamide ,until 36th week (prolonged to 40 or 44 weeks if no smear conversion by end of 16th and 20th week) .
  Interventions: Drug: Bedaquiline; Drug: Pyrazinamide; Drug: Linezolid; Drug: Cycloserine; Drug: Clofazimine

INTERVENTIONS:
Drug: Bedaquiline — 400 mg once daily for 2 weeks then 200mg 3 times per week;
  Other Names: BDQ
Drug: Pyrazinamide — 1500 mg daily
  Other Names: PZA
Drug: Linezolid — 600 mg daily
  Other Names: LZD
Drug: Cycloserine — ≤50kg 500 mg daily, >50kg 750mg daily;
  Other Names: Cs
Drug: Clofazimine — 100 mg daily;
  Other Names: CFZ

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of a combination of bedaquiline, linezolid, cycloserine, clofazimine and pyrazinamide treatments guided by PZA sensitivity for 24 to 36 weeks in subjects with fluoroquinolone-resistant MDR-TB .

DETAILED DESCRIPTION:
The TB-TRUST-plus is a phaseIII, multicenter, open-label trial. The purpose of this study is to assess the feasibility of the ultra-short treatment regimen guided by PZA sensitivity among fluoroquinolone-resistant MDR-TB patients.A total of 200 participants with MDR-TB will be recruited and followed up until 84 weeks after the treatment initiation.

This regimen consists of two periods of 24-36 weeks. During the first 4-8 weeks(waiting for pyrazinamide drug sensitivity test), the regimen consists of bedaquiline, linezolid, cycloserine, clofazimine and pyrazinamide. Then based on molecular PZA drug sensitivity results, patients will be in divided into 3 sub-groups: pyrazinamide-susceptible (PZA-S) patients , pyrazinamide-resistant (PZA-R) patients and pyrazinamide-unavailable (PZA-U)patients.

The Regimen for PZA-S patients, consisting of bedaquiline, linezolid, cycloserine and pyrazinamide, are given until the 24th week (prolonged to 28 or 32 weeks if no smear conversion by end of 16th and 20th week).

PZA-R sub-group regimen, consisting of bedaquiline, linezolid, cycloserine and clofazimine ,are given until 36th week (prolonged to 40 or 44 weeks if no smear conversion by end of 16th and 20th week) .

PZA-U sub-group continue the previous regimen, consisting of bedaquiline, linezolid, cycloserine , clofazimine and pyrazinamide ,until 36th week (prolonged to 40 or 44 weeks if no smear conversion by end of 16th and 20th week) .

The primary objective is to access the treatment success rate without relapse of the PZA sensitivity guided ultra short regimen.

The secondary objective is to access the median time to sputum culture conversion. Safety evaluations performed are the routine lab tests, blood glucose, vital signs, electrocardiograph (ECG), reporting of adverse events, peripheral neuropathy brief examining with the use of a Brief Peripheral Neuropathy rating scale(BPNS) and ophthalmologic examination, including assessment of visual acuity and color vision，physical examinations and chest CT. Adverse events will be monitored and promptly managed during the whole treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in trial treatment and follow-up and can give informed consent
* 18-70 years old
* Has smear-positive pulmonary tuberculosis with initial laboratory results with resistance to rifampicin and isoniazide confirmed by GeneXpert
* documented resistance to fluoroquinolones at screening
* Can use bedaquiline, linezolid, cycloserine, clofazimine and pyrazinamide drugs concerning the availability and costs of essential medicines
* Willing to carry out HIV testing.
* If the patient is a non-menopausal woman, agree to use or have used effective contraception during treatment.
* Have an identifiable address and stay in the area during the study period.
* Willing to follow the follow-up study procedure after the follow-up.

Exclusion Criteria:

* Combined extrapulmonary tuberculosis;
* HIV antibody positive and AIDS patients;
* Critically ill patients, and according to the judgment of the research physician, it is impossible to survive for more than 16 weeks;
* Known to be pregnant or breastfeeding;
* Unable to attend or follow treatment or follow-up time;
* Can not take oral medications;
* Patients with impaired liver function (hepatic encephalopathy, ascites; total bilirubin is more than 2 times higher than the upper limit of normal; ALT or AST is more than 5 times the upper limit of normal);
* Blood muscle spasm is more than 1.5 times the upper limit of normal;
* The investigator believes that there are any social or medical conditions that expose the subject to a safety hazard;
* Simultaneously apply the drugs (glucocorticoids, interferons) that affect the efficacy of this study; and apply the following drugs contraindicated with the study drug, including non-steroidal anti-inflammatory drugs, monoamine oxidase inhibitors (phenethyl hydrazine, different Carbofurs et al), direct or indirect sympathomimetic drugs (such as pseudoephedrine), vasopressor drugs (such as adrenaline, norepinephrine), dopamine drugs (such as dopamine, dobutamine), 5 a serotonin reuptake inhibitor, a tricyclic antidepressant, a serotonin 5-HTI receptor antagonist (amitriptyline), meperidine or buspirone.
* Being allergic or intolerant of any study drug;
* Currently participating in another drug clinical trial;
* QTc interval ≥ 500 milliseconds during screening;
* Hemoglobin is less than 90g/L or platelet is less than 75*10^9/L;
* Have epilepsy, severe depression, irritability or psychosis；
* Alcohol abuse（drinking more than 64g of ethanol a day for male, 42g for female）.
* Subjects receive more than 2 weeks of bedaquiline, linezolid, cycloserine, clofazimine or pyrazinamide 3 months prior to enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Treatment success rate | 84 weeks after the treatment initiation
  To access the treatment success rate without relapse .Treatment outcomes will be classified into favourable outcome and unfavourable outcome.

SECONDARY OUTCOMES:
The median time to Sputum Culture Conversion | Time Frame: 12-36 weeks after treatment initiation
  time from treatment initiation to the first of two consecutive negative sputum cultures without an intervening positive culture in liquid media
The frequency of grade 3 or greater adverse events among patients | 84 weeks after treatment initiation
  to access the proportion of patients who experience grade 3 or greater adverse events (graded according to the Division of AIDS severity criteria for adverse events) during treatment or follow-up;

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PhD, Principal Investigator — Huashan Hospital
Locations (15):
- China (15):
  - The Third People's Hospital of Shenzhen City, Shenzhen, Guangzhou
  - Guiyang Public Health Treatment Center, Guizhou, Guizhou
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Hunan Chest Hospital, Changsha, Hunan
  - Huaihua first people's Hospital, Huaihua, Hunan
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Tuberculosis Control Institute, Xi’an, Shanxi
  - Chest Hospitalof Xinjiang Uygur Autonomous Region of PRC, Ürümqi, Xinjiang
  - Baoshan People's Hospital, Baoshan, Yunnan
  - Yunnan Provincial Infectious Disease Hospital, Kunming, Yunnan
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - Hwa Mei Hosptal,University of Chinese Academy of Sciences(Ningbo No.2 Hospital), Ningbo, Zhejiang
  - Taizhou Enze medical center Enze Hospital, Taizhou, Zhejiang
  - The Central Hospital of Wenzhou City, Wenzhou, Zhejiang
  - Jiangxi Chest Hospital, Nanchang

IPD SHARING:
Plan to Share IPD: No